CLINICAL TRIAL: NCT04471597
Title: Topical Bupivacaine Effect On The Response To Awake Extubation During Emergence From General Anesthesia In Patients Undergoing Elective Thyroidectomy. A Randomized Controlled Study
Brief Title: Topical Bupivacaine Effect On The Response To Awake Extubation During Emergence From General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, principal investigator, lecturer, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6201//12-7-2020
Record Dates: First submitted 2020-07-12; First posted 2020-07-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Thyroid Diseases
Keywords: topical bupivacaine; awake extubation; thyroidectomy; general anesthesia
MeSH Terms: conditions — Thyroid Diseases | interventions — Saline Solution; Bupivacaine

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into two equal groups
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded ( patient and outcome assessors)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): patients will receive 5ml of normal saline 0.9% topically 15 min before the expected end of surgery.
  Interventions: Drug: normal saline 0.9%
- bupivacaine group (Active Comparator): patients will receive 5ml of bupivacaine 0.5% topically 15 min before the expected end of surgery.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: normal saline 0.9% — 5ml of normal saline 0.9% topically 15 min will be installed topically around the ETT using ordinary syringe before the expected end of the surgery, this will be followed by manual ventilation using about the double tidal volume for 6-8 times or more to get air bubbles distributed within the upper airway to anesthetize the oropharynx and spread around ETT to the adjacent mucosal structures (laryngopharynx, larynx, and upper part of the trachea) then the cuff will be inflated to the previous pressure and the patient will be mechanically ventilated as usual.
  Arms: Control group
Drug: Bupivacaine Hydrochloride — 5 ml of bupivacaine 0.5% will be installed topically around the ETT using ordinary syringe before the expected end of the surgery, this will be followed by manual ventilation using about the double tidal volume for 6-8 times or more to get air bubbles distributed within the upper airway to anesthetize the oropharynx and spread around ETT to the adjacent mucosal structures (laryngopharynx, larynx, and upper part of the trachea) then the cuff will be inflated to the previous pressure and patient will be mechanically ventilated as usual.
  Arms: bupivacaine group

SUMMARY:
* Emergence from general anesthesia is often complicated by the ETT-induced emergence phenomena (EP), which include coughing, sympathetic stimulation, sore throat, increased bleeding from the surgical site, and increased intracranial and intraocular pressures.
* Techniques that have been used to help diminish coughing during emergence include "deep" extubation (removal of the endotracheal tube [ETT] while the patient is still in a deep plane of general anesthesia), administration of intravenous (IV) narcotics, or administration of IV lidocaine prior to emergence since systemic narcotics and lidocaine have antitussive properties. However, each of these techniques has limitations. A reliable technique for improving ETT tolerance while facilitating rapid and full emergence from general anesthesia would be desirable in many situations.
* Topical application of bupivacaine to the pharyngeal, laryngeal, and tracheal mucosa will attenuate or even abolish coughing as well as a hemodynamic response during extubation, thus result in increasing the patient's comfort and avoiding potential complications of extubation process.
* Up to the investigator's knowledge there is no study done to evaluate the effect of topical bupivacaine on the incidence of coughing and hemodynamic response during emergence from general anesthesia in patients undergoing elective thyroidectomy.

DETAILED DESCRIPTION:
The process of manipulation of the airway during laryngoscopy, endotracheal intubation, and extubation is usually associated with exaggerated hemodynamic response including tachycardia, hypertension as well as increase intraocular and intracranial pressure[1,2]. The exact mechanism to these hemodynamic responses may be due to the release of catecholamine in the blood by stimulating the sympathetic nervous system during these stressful periods. Acute hemodynamic changes during extubation may lead to life-threatening myocardial ischemia, arrhythmias, pulmonary edema, acute heart failure, or cerebrovascular hemorrhage in high-risk patients and this can increase morbidity and mortality of the patients [3].

Respiratory complications after tracheal extubation are three times more common than induction of anesthesia and intubation [4], as intratracheal tube induces laryngeal irritation that transmitted through rapidly acting receptors which are located throughout the trachea, involved in the cough reflex and subsequently lead to coughing and bucking that frequently occur during extubation and may lead to negative pressure pulmonary edema as well as, laryngeal edema and sore throat [5, 6].

Various techniques have been applied to attenuate the hemodynamic responses and coughing during emergence and extubation. They include deep extubation, administration of intravenous (IV) short-acting narcotics, calcium channel blockers, and dexmedetomidine [7,8], as well as lidocaine which is considered one of the commonly used drugs either through IV route, endotracheal tube (ETT) cuff, or laryngotracheal route[1,9]. Concern about the use of these drugs includes respiratory depression, delayed emergence from anesthesia, postoperative nausea and vomiting, sedative effects, and short action time [10].

Bupivacaine is a kind of sodium channel blocker local anesthetics used as topical anesthesia that suppresses cough by inhibiting the progression of the action potential in the tracheal touch-sensitive Aδ fibers (cough receptors)[10]. The plasma protein binding of bupivacaine exceeds 90%, whereas lidocaine protein binding is 65- 75%, [11] and it is well known that the duration of local anesthetics is influenced by their protein binding characteristics, as the affinity for plasma proteins corresponds to the affinity for protein binding at the sodium channel receptor site, that results in prolongation of the presence of the anesthetic effect at the site of action [12, 13].

the investigators hypothesize that usage of topical bupivacaine may have an impact on decreasing incidence of coughing and alleviating hemodynamic response during awake extubation and emergence from general anesthesia in post-thyroidectomy patients.

ELIGIBILITY:
Inclusion Criteria:

Patient acceptance. BMI < 35kg/m2. ASA I and ASA II. Scheduled for elective thyroidectomy under general anesthesia

Exclusion Criteria:

Patient refusal. History or anticipated difficult intubation. Chronic respiratory disease such as chronic obstructive pulmonary disease or asthma.

Recent respiratory tract infection in the last month, chronic cough, and current smoking.

History of laryngeal or tracheal surgery or pathology. Patients with symptomatic gastric reflux. Patients with a known history of allergy to study drugs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Grade of coughing | procedure (measured within the extubation time)
  will be assessed as Grade 0: no cough; Grade 1: single cough with mild severity; Grade 2: cough lasting less than 5 s with moderate severity; Grade 3: sustained bouts of persistent cough more than 5 s.

SECONDARY OUTCOMES:
oxygen saturation(SpO2) | will be recorded at base line, after administration of the study drug, before extubation, then at 1 min, 2min, 5min, and 10 min immediately following extubation.
heart rate | will be recorded at base line, after administration of the study drug, before extubation, then at 1 min, 2min, 5min, and 10 min immediately following extubation.
  Hemodynamics
mean arterial blood pressure | will be recorded at base line, after administration of the study drug, before extubation, then at 1 min, 2min, 5min, and 10 min immediately following extubation.
  Hemodynamics
Extubation time | Procedure -from the end of the anesthesia (discontinuation of isoflurane) to the time the endotracheal tube will be pulled out
  removal of the endotracheal tube [ETT] while the patient is still in a deep plane of general anesthesia
Sore throat degree | 1 , 2 , 4, 6 and 12 hours postoperatively.
  will be assessed by visual analogue scale (VAS) scale, On a scale of 0-10, the patient will learn to quantify postoperative sore throat pain where 0= No pain and 10= Maximum worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Shabnum T, Ali Z, Naqash IA, Mir AH, Azhar K, Zahoor SA, Mir AW. Effects of Lignocaine Administered Intravenously or Intratracheally on Airway and Hemodynamic Responses during Emergence and Extubation in Patients Undergoing Elective Craniotomies in Supine Position. Anesth Essays Res. 2017 Jan-Mar;11(1):216-222. doi: 10.4103/0259-1162.200239. PMID 28298788
- [Background] Meng YF, Cui GX, Gao W, Li ZW. Local airway anesthesia attenuates hemodynamic responses to intubation and extubation in hypertensive surgical patients. Med Sci Monit. 2014 Aug 26;20:1518-24. doi: 10.12659/MSM.890703. PMID 25175842
- [Background] Fang P, Zong Z, Lu Y, Han X, Liu X. Effect of topical ropivacaine on the response to endotracheal tube during emergence from general anesthesia: a prospective randomized double-blind controlled study. BMC Anesthesiol. 2018 Sep 27;18(1):134. doi: 10.1186/s12871-018-0601-x. PMID 30261837
- [Background] Phero JC, Prithvi Raj P, Knarr D, Turner P, Denson DD, Vigdorth E, Edstrom HH. Absorption of bupivacaine after topical application to the oropharynx. Anesth Prog. 1987 Sep-Oct;34(5):187-90. PMID 3479919
- [Background] Mogensen S, Sverrisdottir E, Sveinsdottir K, Treldal C, Jensen K, Jensen AB, Kristensen CA, Jacobsen J, Kreilgaard M, Petersen J, Andersen O. Absorption of Bupivacaine after Administration of a Lozenge as Topical Treatment for Pain from Oral Mucositis. Basic Clin Pharmacol Toxicol. 2017 Jan;120(1):71-78. doi: 10.1111/bcpt.12644. Epub 2016 Sep 26. PMID 27430990
- [Background] Fisman EZ, Shapira I, Motro M, Pines A, Tenenbaum A. The combined cough frequency/severity scoring: a new approach to cough evaluation in clinical settings. J Med. 2001;32(3-4):181-7. PMID 11563816